CLINICAL TRIAL: NCT00465192
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study Comparing the Efficacy and Safety of 17-Beta Estradiol 10 Micrograms and 25 Micrograms (Vagifem) Doses in Treatment of Estrogen Deficiency-Derived Atrophic Vaginitis
Brief Title: Efficacy and Safety of 17-Beta Estradiol in Treatment of Atrophic Vaginitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VAG/PD/009/USA
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Menopause; Postmenopausal Vaginal Atrophy
MeSH Terms: interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: estradiol, 10 mcg
Drug: estradiol, 25 mcg
Drug: placebo

SUMMARY:
This trial was conducted in the United States of America (USA). This trial aimed for a comparison between the effect of two different doses of estradiol on parameters related to efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy
* Postmenopausal
* Hysterectomized or non-hysterectomized
* Moderate or severe vaginal dryness and soreness

Exclusion Criteria:

* Known, suspected, or past history of breast cancer
* Known, suspected, or past history of hormone-dependent tumor
* Genital bleeding of unknown etiology
* Acute thrombophlebitis or thromboembolic disorders or a past history of these conditions, associated with previous estrogen use
* Vaginal infection
* Use of exogenous corticosteroids or sex hormones within 8 weeks of starting active treatment in study
* Use of vaginal, oral or vulvar homeopathic preparations within seven days of starting active treatment in study
* History of treatment with diethylstilbestrol

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 1994-08-31 (Actual); Primary Completion 1995-11-30 (Actual); Study Completion 1995-11-30 (Actual)

PRIMARY OUTCOMES:
Relief of vaginal symptoms | following 12 weeks of treatment.

SECONDARY OUTCOMES:
Adverse events
Hematology and chemisty tests, and endometrial biopsy
Vaginal and urethral cytology, and grading of vaginal health

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S

REFERENCES:
- [Derived] Bachmann G, Lobo RA, Gut R, Nachtigall L, Notelovitz M. Efficacy of low-dose estradiol vaginal tablets in the treatment of atrophic vaginitis: a randomized controlled trial. Obstet Gynecol. 2008 Jan;111(1):67-76. doi: 10.1097/01.AOG.0000296714.12226.0f. PMID 18165394
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com